CLINICAL TRIAL: NCT05761496
Title: Metal and Plastic Biliary Stents to Drain Malignant Distal Biliary Strictures. Registry of the Italian Society of Digestive Endoscopy.
Brief Title: Metal and Plastic Biliary Stents to Drain Malignant Distal Biliary Strictures.
Acronym: PROTESIED
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Tringali Andrea, MD, PhD, Assitant Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2767
Record Dates: First submitted 2023-02-25; First posted 2023-03-09 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Biliary Stricture; Stent Stenosis
Keywords: Biliary stricture; Plastic stent; Self Expandable Metal stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Biliary stents insertion — Endoscopic placement of plastic and metal biliary stents

SUMMARY:
Multicentric Italian registry aimed to evaluated the role and results of plastic and metal stents in the treatment of malignant distal biliary strictures

ELIGIBILITY:
Inclusion Criteria:

* Malignant distal biliary stricture
* Need for Palliative and pre-operative biliary drainage
* Age > 18
* Signature of the informed consent

Exclusion Criteria:

* Previous endoscopic/radiological biliary drainage
* Stricture close to the main hepatic confluence(< 2 cm)
* Duodenal stenosis
* Post- surgical altered anatomy
* Benign disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring for the first time drainage of malignant distal biliary stricture
Sampling Method: Non-Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the potency of biliary stents (plastic and metal) | through study completion, an average of 1 year
  Time to occurrence of jaundice/cholangitis

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tringali, MD, PhD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS, Rome, Italy
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy